CLINICAL TRIAL: NCT07185334
Title: Single-Stage Prepectoral Placement of Textured Implants Using a Polyester Mesh Endoprostheses With Fluoropolymer Coating in Patients With Breast Cancer
Acronym: FluoropolyMesh
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Laisan Shaikhelislamova, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50
Record Dates: First submitted 2025-09-02; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Reconstruction; Coated Materials; Reconstruction Breast Surgery; MASH With Fibrosis
Keywords: Fluoropolymer coated mesh; Implant-based reconstruction in breast cancer patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Intervention Model Description: Main group- The main group will consist of patients undergoing surgical treatment for subcutaneous mastectomy using a polyester mesh endoprosthesis with a fluoropolymer coating, with simultaneous prepectoral placement of textured implants.
  Control group-The control group will consist of patients who undergo surgical treatment for subcutaneous mastectomy, with simultaneous placement of textured breast implants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main group (Experimental): The main group will consist of patients with the planned volume of surgical intervention: subcutaneous mastectomy using a polyester mesh endoprosthesis with a fluoropolymer coating and simultaneous prepectoral placement of textured implants.
  Interventions: Procedure: Subcutaneous mastectomy using a fluoropolymer-coated polyester mesh endoprosthesis with simultaneous prepectoral placement of textured implants.
- Control group (Other): The control group will consist of patients who undergo surgical treatment for subcutaneous mastectomy, with simultaneous placement of textured breast implants with no polyester mesh endoprosthesis with a fluoropolymer coating
  Interventions: Procedure: Subcutaneous mastectomy with simultaneous prepectoral placement of textured implants.

INTERVENTIONS:
Procedure: Subcutaneous mastectomy using a fluoropolymer-coated polyester mesh endoprosthesis with simultaneous prepectoral placement of textured implants. — For this group of patients, the planned volume of surgical intervention is: subcutaneous mastectomy using a polyester mesh endoprosthesis with a fluoropolymer coating and one-stage prepectoral installation of textured implants.
  Arms: Main group
Procedure: Subcutaneous mastectomy with simultaneous prepectoral placement of textured implants. — This group of patients will undergo surgical intervention in deep subcutaneous mastectomy with simultaneous prepectoral placement of textured implants.
  Arms: Control group

SUMMARY:
This study aims to evaluate the efficacy of using a polyester mesh endoprosthesis with a fluoropolymer coating in reducing postoperative complications, particularly protrusions, following subcutaneous mastectomy with simultaneous prepectoral placement of textured breast implants in women with breast cancer

DETAILED DESCRIPTION:
The study includes female patients aged 18 and above with a verified breast cancer diagnosis, ECOG performance status 0-1, and clinical stage T1-T3, N0-3, M0, who provide informed consent. Exclusion criteria involve intolerance or allergic reactions to mesh endoprostheses or implants and a subcutaneous adipose tissue thickness of less than 5 mm (measured via Pinch Test). Participants will be non-randomly allocated into two groups: the main group, receiving a polyester mesh endoprosthesis with fluoropolymer coating alongside textured implants, and the control group, receiving textured implants alone. Surgical procedures will involve subcutaneous mastectomy with implant placement based on preoperative measurements of breast dimensions, with or without nipple-areolar complex preservation. Postoperative follow-ups at 1, 3-6, and 9-12 months will assess complications such as protrusions, seromas, implant contouring (rippling), capsular contracture, and dystopia via physical examination and ultrasound. The hypothesis posits that the use of mesh endoprostheses will lower protrusion rates compared to standard implant placement, offering a potential advancement in reducing postoperative risks in breast reconstruction for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a verified breast cancer diagnosis over 18 years of age;
2. ECOG 0-1;
3. Stage: clinical T1, T2 or T3, N0-3, M0;
4. The thickness of subcutaneous adipose tissue (Pinch Test) is more than 5 mm
5. Signed informed voluntary consent.

Exclusion Criteria:

1. Women under 18 years of age;
2. ECOG 2-4;
3. Stage: clinical T4, M1;
4. The thickness of subcutaneous adipose tissue (Pinch Test) is less than 5 mm;
5. Intolerance and / or allergic reaction to the mesh endoprosthesis, implant and/or its component;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of protrusions throughout the year | 1 year
  Implant protrusion is a complication that occurs after reconstructive plastic surgery. In this type of surgery, the implant is displaced from its anatomically correct position leading to its protrusion through the skin. This happens when the integrity or strength of the tissues that hold the implant (such as capsules, muscles, and fascia) is compromised.

SECONDARY OUTCOMES:
1. Frequency of seroma 2. Frequency of Rippling 3. Frequency of Capsular contracture 4. Frequency of Dystopia | 1 year
  1. Seroma is a pathological accumulation of serous fluid in the tissues after surgery or trauma. Most often, this condition develops after operations that affect large areas of the skin and subcutaneous fat.
  2. Rippling - represents contouring of the implant through the surface of the mammary glands, expressed by folds in the area of implantplacement.Sometimes it is called "skin ripples" or"washboard effect".
  3. Capsular contracture is the formation of connective tissue around the implant, resulting in compression and deformation of the prosthesis.
  4. Dystopia is a displacement of the implant relative to its original correct anatomical position, which leads to breast deformity, asymmetry, or functional discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No